CLINICAL TRIAL: NCT00756847
Title: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of XL147 (SAR245408) in Combination With Paclitaxel and Carboplatin in Subjects With Solid Tumors
Brief Title: Safety Study of XL147 (SAR245408), in Combination With Paclitaxel and Carboplatin in Adults With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11435; XL147-003 (Other: (Other study code))
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Cancer; Non-Small Cell Lung Cancer; Endometrial Carcinoma; Ovarian Carcinoma
Keywords: Solid Tumors; NSCLC; Ovarian Cancer; Endometrial Cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Endometrial Neoplasms; Ovarian Neoplasms | interventions — XL147; Paclitaxel; Carboplatin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: XL147 (SAR245408),; Drug: paclitaxel; Drug: carboplatin

INTERVENTIONS:
Drug: XL147 (SAR245408), — Gelatin capsules supplied in 25- and 100-mg strengths; daily dosing
Drug: paclitaxel — Intravenous injection dosed once every three weeks
  Other Names: Taxol®
Drug: carboplatin — Intravenous injection dosed once every three weeks

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of XL147 in combination with paclitaxel and carboplatin in adults with solid tumors. XL147 is a new chemical entity that inhibits PI3 Kinase. Inactivation of PI3K has been shown to inhibit growth and induce apoptosis (programmed cell death) in tumor cells. In clinical practice, the combination of paclitaxel and carboplatin is an accepted treatment regimen for various solid tumors, including ovarian cancer, endometrial cancer and non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of:

  * Advanced solid tumor that is no longer responding to therapies OR
  * Advanced or recurrent endometrial carcinoma OR
  * Advanced or recurrent ovarian carcinoma OR
  * Unresectable (Stage IIIB or IV) NSCLC
* ECOG Performance Status 0-1 (ECOG status of 2 may be considered following discussion and agreement with sponsor)
* Adequate organ and bone marrow function as defined by hematological and serum chemistry limits
* At least 18 years old
* Both men and women must practice adequate contraception
* Informed consent

Exclusion Criteria:

* Restriction of some therapies/medications within specific timeframes prior to enrollment and during the study including prior therapy with PI3K, AKT, or mTOR inhibitors, cytotoxic chemotherapy, biologic agents, nitrosoureas or mitomycin C, small-molecule kinase inhibitors, non-cytotoxic hormonal agents
* Known allergy or hypersensitivity to any of the components of the treatment formulations
* Taking oral corticosteroids chronically or > 1 mg/day warfarin
* Not recovered from the toxic effects of prior therapy
* History of diabetes mellitus.
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding
* Congestive heart failure, unstable angina, or a myocardial infarction within 3 months of entering the study.
* HIV positive
* Diagnosis of another malignancy may exclude subject from study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, and MTD of XL147 administered in combination with paclitaxel (at doses up to 175 mg/m2) and carboplatin in subjects with advanced solid tumors | Assessed at periodic visits
To evaluate the safety, tolerability, and MTD of XL147 administered in combination with paclitaxel (at doses up to 225 mg/m2) and carboplatin in subjects with NSCLC | Assessed at periodic visits

SECONDARY OUTCOMES:
To investigate the relationship between selected biomarkers and efficacy and safety outcomes | Assessed at periodic visits
To assess plasma pharmacokinetics (PK) of XL147, paclitaxel, and carboplatin when used in combination | Assessed at periodic visits
To evaluate preliminary antitumor activity of XL147 in combination with carboplatin and paclitaxel | Assessed at periodic visits

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (4):
  - Investigational Site Number, St Louis, Missouri
  - Investigational Site Number, Oklahoma City, Oklahoma
  - Investigational Site Number, Houston, Texas
  - Investigational Site Number, Madison, Wisconsin

REFERENCES:
- [Derived] Wheler J, Mutch D, Lager J, Castell C, Liu L, Jiang J, Traynor AM. Phase I Dose-Escalation Study of Pilaralisib (SAR245408, XL147) in Combination with Paclitaxel and Carboplatin in Patients with Solid Tumors. Oncologist. 2017 Apr;22(4):377-e37. doi: 10.1634/theoncologist.2016-0257. Epub 2017 Mar 8. PMID 28275119